CLINICAL TRIAL: NCT00728260
Title: Post-licensure Safety Surveillance Study of Routine Use of Meningococcal (Groups A, C, Y, and W-135) Polysaccharide Diphtheria Toxoid Conjugate Vaccine (Menactra®) in Recipients 2 to 10 Years of Age.
Brief Title: 36-Month Post-marketing Surveillance and Analysis of Menactra Vaccine in 2-10 Year Olds
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: MTA38
Record Dates: First submitted 2008-05-07; First posted 2008-08-05 (Estimated); Results first posted 2015-02-12 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-02

CONDITIONS: Meningitis; Meningococcal Disease
Keywords: Meningitis; Meningococcal disease; Menactra vaccine
MeSH Terms: conditions — Meningitis; Meningococcal Infections

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Menactra Vaccine Recipients: Children 2 years through 10 years of age who received Menactra vaccine within Kaiser Permanente during the study period. They served as their own controls for evaluation of acute (Days 0-30) events. Rates of events occurring during Days 0-30 following vaccination were compared to rates of events occurring during Days 31-60 following vaccination.
  Six-month surveillance: For each individual receiving Menactra vaccine, the rate of an event in the 30-day follow-up period was compared with the rate of the same event in the 31-180-day follow-up period using age, sex, and seasonality as covariates in Cox regression analyses.
  Menactra vaccine was administered according to routine clinical practice.
  Interventions: Biological: None administered in this study

INTERVENTIONS:
Biological: None administered in this study — N/A in this study

SUMMARY:
To further characterize the safety profile of Menactra vaccine and to identify any signals of potentially vaccine-related adverse events (AEs) not detected during pre-licensure studies.

ELIGIBILITY:
Inclusion Criteria:

* Receipt of Menactra vaccine during the study period.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Past receipt of Menactra vaccine
Sampling Method: Non-Probability Sample
Enrollment: 1421 (Actual)
Dates: Start 2005-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (1):
- Oakland, California, United States

REFERENCES:
- [Derived] Hansen J, Zhang L, Eaton A, Baxter R, Robertson CA, Decker MD, Greenberg DP, Bassily E, Klein NP. Post-licensure safety surveillance study of routine use of quadrivalent meningococcal diphtheria toxoid conjugate vaccine (MenACWY-D) in infants and children. Vaccine. 2018 Apr 12;36(16):2133-2138. doi: 10.1016/j.vaccine.2018.02.107. Epub 2018 Mar 14. PMID 29550195
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participant accrual occurred from 18 October 2007 through 17 October 2010. Kaiser Permanente databases were reviewed for this study.
Pre-assignment Details: Medical utilization databases were reviewed for children 2 through 10 years of age receiving Menactra vaccine within Kaiser Permanente to identify the following medical care events during the 6 months after Menactra vaccination: all outcomes from hospitalizations and emergency department visits and selected outcomes from clinic visits.
Period: Overall Study
Arm/Group | Menactra Vaccine Recipients
Started | 1421
Completed | 1421
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Children 2 through 10 years of age who received Menactra vaccine within Kaiser Permanente during the study period.
Arm/Group | Menactra Vaccine Recipients
Number analyzed (Participants) | 1421
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1421
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.36 (2.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 709
  Male | 712
Region of Enrollment [Number; unit: participants]
  United States | 1421
Seasonality [Number; unit: Participants] — Data represent participants receiving vaccine during each time period shown. One participant had received more than one dose of Menactra vaccine; each dose is counted in the seasonality section.
  Participants
    December - February | 163
    March - May | 372
    June - August | 593
    September - November | 294
Indication for Vaccination [Number; unit: Participants] — Based on automated subject data. Participants may be included in more than 1 category
  Participants
    Asplenia (Surgical or Congenital) | 17
    Complement Deficiency | 2
    Hereditary Elliptocytosis | 1
    Hereditary Spherocytosis | 8
    Sickle Cell Disease | 44
    Thalassemias | 22
    Other Hemoglobinopathy | 9
    Human Immunodeficiency Virus Infection | 1
    Travel-Related | 364
    Not Available | 987

OUTCOME MEASURES:

1. Primary Outcome: Summary of Diagnoses With Elevated Findings for Risk-Window vs. Control-Window Comparisons at the 5% Significance Level.
Description: Incidence rates for each diagnosis were calculated as the number of events divided by person-time and expressed as events per 1,000 person-months in each comparison window. Clinical setting is given in parenthesis as (H) for hospital.
Time Frame: Day 0 up to Day 30 post-vaccination
Population: All persons who received Menactra vaccine during the study period were included in the analysis.
Measure: Number; unit: Events per 1,000 person-months
Arm/Group | Menactra Vaccine Recipients
Number analyzed (Participants) | 1421
Events per 1,000 person-months
  Cellulitis and abscess (All ages combined; H) | 1.4
  Cellulitis and abscess (Subj.10 Yrs Old; H; n=870) | 2.3

2. Other Pre Specified Outcome: Rates of Serious Adverse Events Per 1000 Doses at During 6 Months After Menactra Vaccination From Inpatient Database - All Ages Combined
Description: Only persons who received Menactra vaccine during the study period were surveyed and included in this outcome.
Time Frame: Day 0 up to 6 months post-vaccination
Population: Only persons who received Menactra vaccine during the study period were included in the analysis.
Measure: Number; unit: Events per 1,000 doses
Arm/Group | Menactra Vaccine Recipients
Number analyzed (Participants) | 1421
Events per 1,000 doses
  Abdominal pain | 0.70
  Aspergillosis | 0.70
  Asthma | 0.70
  Cellulitis and abscess | 1.41
  Cerebral palsy | 0.70
  Congenital anomaly of ureter | 0.70
  Congenital atresia | 0.70
  Digestive congenital anomalies | 070
  Febrile illness | 2.81
  Feeding problem | 0.70
  Hereditary spherocytosis | 0.70
  Hydronephrosis | 0.70
  Malignant neoplasm | 5.63
  Other non-traumatic joint disorders | 0.70
  Pneumonia | 0.70
  Psychiatric | 0.70
  Pyogenic arthritis | 0.70
  Respiratory infection, upper | 0.70
  Sickle cell anemia | 5.63
  Small bowel obstruction | 0.70
  Trauma | 2.11

3. Primary Outcome: Summary of Diagnoses With Elevated Findings for Risk-Window vs. Control-Window Comparisons at the 5% Significance Level.
Description: as for outcome 1
Time Frame: Day 31 up to Day 180 post-vaccination
Population: All persons who received Menactra vaccine during the study period were included in the analysis.
Measure: Number; unit: Events per 1,000 person-months
Arm/Group | Menactra Vaccine Recipients
Number analyzed (Participants) | 1421
Events per 1,000 person-months
  Cellulitis and abscess (All ages combined; H) | 0.0
  Cellulitis and abscess (Subj.10 Yrs Old; H; n=870) | 0.0

ADVERSE EVENTS:
Time Frame: Surveillance period for serious adverse events was from the day of vaccination up to 6 months post-vaccination from the inpatient database.
Arm/Group | Menactra Vaccine Recipients
Serious Adverse Events (participants affected / at risk) | 16/1421
Other Adverse Events (participants affected / at risk) | 0/1421
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Menactra Vaccine Recipients (N=1421)
Congenital Anomaly of ureter (Congenital, familial and genetic disorders) | 1
Sickle Cell Anemia (Congenital, familial and genetic disorders) | 8
Abdominal Pain (Gastrointestinal disorders) | 1
Febrile Illness (General disorders) | 4
Feeding problem (Metabolism and nutrition disorders) | 1
Aspergillosis (Infections and infestations) | 1
Pyogenic arthritis (Infections and infestations) | 1
Respiratory infection, upper (Infections and infestations) | 1
Trauma (Injury, poisoning and procedural complications) | 3
Psychiatric (Psychiatric disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Small bowel obstruction (Gastrointestinal disorders) | 1
Digestive congenital anomalies (Congenital, familial and genetic disorders) | 1
Congenital atresia (Congenital, familial and genetic disorders) | 1
Cerebral palsy (Congenital, familial and genetic disorders) | 1
Cellulitis and abscess (Infections and infestations) | 2
Hereditary spherocytosis (Congenital, familial and genetic disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Malignant neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
Other non-traumatic joint disorders (Musculoskeletal and connective tissue disorders) | 1
Pneumonia (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.